CLINICAL TRIAL: NCT00511498
Title: Effect of Nightly Versus Prn Sildenafil on Early Return of Erectile Function Following Nerve-Sparing Laparoscopic Radical Prostatectomy
Brief Title: Effect of Nightly Versus Prn Sildenafil on Early Return of Erectile Function Following Laparoscopic Radical Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Christian Pavlovich, M.D., Johns Hopkins University
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: NA_00001428
Record Dates: First submitted 2007-08-03; First posted 2007-08-06 (Estimated); Last update posted 2008-12-01 (Estimated); Status verified 2008-11

CONDITIONS: Prostate Cancer
Keywords: Laparoscopic Radical Prostatectomy; Nightly sildenafil
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Arm (Placebo Comparator): Placebo nightly
  Interventions: Drug: Sildenafil
- Drug (Active Comparator): Sildenafil 50mg nightly
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil — 50 mg daily at bedtime
  Other Names: Viagra

SUMMARY:
The ability of sildenafil to aid in the return of erections after nerve-sparing radical prostatectomy has been established. Patients who had either one or both neurovascular bundles spared demonstrated dramatically better responses to "as needed" sildenafil than those that did not, and a positive erectile response to sildenafil was only seen in patients in whom at least one NVB was spared. This study has been designed to determine if sildenafil taken nightly works better than sildenafil on as "as needed" basis for the return of erectile function. The investigators hypothesis is that sildenafil taken nightly promotes a more rapid return of erectile function after nerve-sparing laparoscopic radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Male sex
2. Age < 65
3. IIEF erectile function domain score > 26 (out of 30 points possible for this subscale)
4. Steady sexual partner
5. Untreated prostate cancer TNM stage < cT2bNxMx (cT1a, cT1b, cT1c, cT2a) and Gleason grade < 8.
6. Willingness to participate in a clinical trial as manifested by informed consent
7. Actually undergo nerve-sparing LRP surgery

Exclusion Criteria:

1. Not fulfilling all of the criteria for entry above
2. Any prior prostate cancer treatment (radiation, hormonal deprivation, chemotherapy)
3. Contraindication to sildenafil (e.g. nitrates, hypersensitivity)
4. Existing PDE5 inhibitor requirement for functional erection (e.g. for intercourse) preoperatively
5. Obstructive sleep apnea

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2006-03; Primary Completion 2007-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
IIEF score | 13 months

CONTACTS AND LOCATIONS:
Overall Officials: Christian P Pavlovich, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States